CLINICAL TRIAL: NCT04687891
Title: Transabdominal Versus Transvaginal Ultrasound to Assess the Thickness of the Lower Uterine Segment at Term in Women With Previous One Cesarean Section.
Brief Title: Transabdominal Versus Transvaginal Ultrasound to Assess the Thickness of the Lower Uterine Segment.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, Principal Investigator, Cairo University
Other Study IDs: 35/2020
Record Dates: First submitted 2020-12-24; First posted 2020-12-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Trans Abdominal Ultrasound; Transvaginal Ultrasound; Lower Uterine Segment Thickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transabdominal ultrasound and transvaginal ultrasound — Within a week before scheduled delivery,antepartum transabdominal and transvaginal ultrasound will be performed with moderately full bladder.

SUMMARY:
aims to determine the accuracy of measurement of the LUS thickness by trans-abdominal and transvaginal ultrasound at term pregnancy in comparison to the actual thickness of LUS measured with manual caliper measurement during cesarean delivery.

Study hypothesis: In women with previous cesarean delivery, determination of the LUS thickness can be done by trans-abdominal and transvaginal ultrasound at term pregnancy and compared to the actual thickness of LUS measured with a manual caliper at cesarean delivery.

Study question: considering transabdominal & transvaginal ultrasound, which of them would be more accurate in the assessment of LUS thickness?

ELIGIBILITY:
Inclusion Criteria:

* Age (20:40 years old).
* Women at term (37:40 weeks).
* With singleton pregnancy.
* Presenting by vertex (cephalic presentation).
* Having adequate liquor.
* Previous delivered by cesarean delivery one time.

Exclusion Criteria:

* Fetal malformations, e.g fetal hydrops.
* Uterine malformations, e.g bicornuate uterus.
* Placental malformations, e.g placenta praevia, placenta accrete.
* Uterine surgery is other than a cesarean, e.g myomectomy.
* Women in labor (painful, regular uterine contractions, cervical dilatation, tender scar, and discomfort is not stopped by sedation).
* Obese patients (BMI >30 kg/m2)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 130 pregnant women at term with a previous one cesarean section admitted for an elective cesarean delivery will be enrolled. LUS thickness will be measured using both TVS and TAS prior to the cesarean. The actual thickness of the LUS will be measured using a sterile metal ruler before the neonate had been delivered.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
accuracy test for measuring | 1 week
  The accuracy of measurement of the LUS thickness by trans-abdominal and transvaginal ultrasound at term pregnancy in comparison to actual thickness of LUS measured with manual caliper at cesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine - Cairo university, Cairo, Kasr El Ainy, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nagy Afifi A, Ahmed Taymour M, Mamdouh El-Khayat W. Transabdominal versus transvaginal ultrasound to assess the thickness of lower uterine segment at term in women with previous cesarean section. Eur J Obstet Gynecol Reprod Biol. 2022 Apr;271:145-151. doi: 10.1016/j.ejogrb.2022.01.027. Epub 2022 Feb 7. PMID 35203047